CLINICAL TRIAL: NCT06988865
Title: Benign Migratory Glossitis Associated With Antiangiogenic Drugs Used in Cancer Treatment
Brief Title: Benign Migratory Glossitis Associated With Antiangiogenic Drugs
Status: Completed | Type: Observational
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, MAURICIO NEVES GOMES, Assistant, Dental Oncology Service, Instituto do Câncer do Estado de São Paulo (ICESP-FMUSP), Instituto do Cancer do Estado de São Paulo
Other Study IDs: Ethics Committee : 6.901.573
Record Dates: First submitted 2025-05-01; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Geographic Tongue
Keywords: antiangiogenic drugs; glossitis benign migratory
MeSH Terms: conditions — Neoplasms; Glossitis, Benign Migratory

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- angiogenesis inhibitors: Oral clinical manifestation
  Interventions: Other: Clinical evaluation

INTERVENTIONS:
Other: Clinical evaluation — treatment methods, associated symptoms, evolution and clinical presentation
  Other Names: clinical images

SUMMARY:
Oral clinical descriptions related to adverse events in patients treated with those elective multi-targeted receptor tyrosine kinase inhibitors and a recombinant humanised monoclonal antibody

DETAILED DESCRIPTION:
Electronical medical and dental records, high-resolution digital photograph were reviewed. Demographic data, medical background, clinical and laboratory information were recorded for each individual case.

ELIGIBILITY:
Inclusion Criteria:

* patient's charts which underwent antiangiogenic targeted drugs

Exclusion Criteria:

* chemoterapy without angiogenesis inhibitors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital -Instituto do Cancer do Estado de Sao Paulo-ICESP
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-07-16 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Benign migratory glossitis | From enrollment to the end of study at 7 years
  erythematous erosions, with loss of filiform papillae, surrounded by white circinate rims on the dorsal tongue

SECONDARY OUTCOMES:
Adverse events | From enrollment to the end of study at 7 years
  Dysgeusia , dermatologic toxicities such as skin erythemas and vesicles on the palms of the hands and burning sensation

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Neves Gomes, PhD, Principal Investigator — Instituto do Cancer do Estado de São Paulo; Wagner Gomes da Silva, PhD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Cancer do Estado de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
undecided